CLINICAL TRIAL: NCT05345340
Title: Effectiveness of Telemedicine on Health Outcomes (Clinical, Humanistic, Economic) in the Management of Patients With Functional Motor Disorder: Randomised Controlled Clinical Trial
Brief Title: Telemedicine in Functional Motor Disorder
Acronym: TeleFMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Collaborators: Marialuisa Gandolfi (Unknown)
Responsible Party: Principal Investigator, Michele Tinazzi, MD, PhD, Full Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TeleFMD-BRFVr
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Functional Movement Disorder
Keywords: Telemedicine; Gait; Economic costs; Pain; Fatigue
MeSH Terms: conditions — Conversion Disorder; Pain; Fatigue | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: This is a single-blind randomized-controlled trial (RCT) with 2-parallel arms comparing the effects between the experimental group (EG) and control group (CG). After screening, a simple randomization list will be generated by a physician using an automated randomization system (www.randomization.com) (allocation ratio 1:1) to assign eligible patients to either the EG or the CG. Group allocation will be kept concealed.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the type of intervention performed by the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Group (Experimental): Patients will receive an individualized intensive 5-day rehabilitation program (2 hours/day, five days/week, one week) by a qualified physiotherapist at the USD Parkinson's Disease and Movement Disorders Unit of Verona (Italy) followed by an individualized self-management program implemented with the Digital Telemedicine platform support ((PHOEMA G.P.I PLATFORM, GPI spa, Trento, Italy). Telemedicine will consist of 24 tele-sessions (1 h/day, one day/week, 24 weeks) and two self-management sessions (1 h/day, two days/week, 24 weeks). For each patient, the duration of the activity, number of steps taken, distance traveled (km), Kcal consumed, duration of inactivity, total hours of sleep, and number of training sessions performed will be monitored through Polar Vantage M devices.
  Interventions: Other: Telemedicine
- Control Group (Active Comparator): Patients will receive the same individualized intensive 5-day rehabilitation program (2 hours/day, 5 days/week, 1 week) of the Telemedicine Group by a qualified physiotherapist at the USD Parkinson's Disease and Movement Disorders Unit of Verona (Italy) followed by a home-based self-management plan (Treatment, as usual, 1 h/day, 3 days/week, 24 weeks) without any Digital Telemedicine platform support.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Telemedicine — The 5-day rehabilitation program will consist of exercises to re-establish standard movement patterns within a multidisciplinary etiological framework, according to a validated rehabilitation protocol for FMDs. Treatment will be tailored to the needs of each patient, following general treatment principles in physiotherapy for FMDs.
  Telemedicine sessions: the patient will perform specific exercises under the supervision of a qualified physiotherapist to provide feedback on the execution and adapt the treatment according to clinical changes/improvements.
  Polar Vantage M devices will collect the objective measurement after the 5-day rehabilitation program (for five consecutive days), week 12 (for five consecutive days), and week 24 (for five consecutive days).
  Arms: Telemedicine Group
Other: Usual care — The 5-day rehabilitation program will be the same as the telemedicine group. A self-management paper log will be given to the patient at the end of the 5-day rehabilitation program. It will include goals, activity plans, and strategies to be used for retraining movements and redirecting attention. Videos stored on the patients' digital device (i.e., tablet, mobile) will include exercises demonstration and execution and strategies to retrain movements. Patients will be encouraged to perform the self-management plan at home on their own (or with their caregivers' help) which will be reported in a paper log and video recorded. The subjective assessment of the patient's motor activity will be collected by clinical diaries focusing on gait and activity level.
  Arms: Control Group

SUMMARY:
Functional motor disorders (FMDs) are a broad spectrum of functional neurological disorders, referring to abnormal movements like dystonia, tremor, and gait/balance disorders. Patients with FMDs experience high degrees of disability and distress equivalent to those suffering from degenerative neurological diseases. Rehabilitation is essential in managing FMDs. However, the current systems of rehabilitation delivery face two main challenges. Patients are not receiving the amount and kind of evidence-based rehabilitation they need due to the lack of rehabilitation professionals' experts in the field. The rehabilitation setting is not adequate for the long-term management and monitoring of these patients. To date, no randomized controlled trials are evaluating the effectiveness of Telemedicine in the management of patients with FMD. This is a single-blind randomized-controlled trial (RCT) with 2-parallel arms to demonstrate the effectiveness and superiority of a 5-day intensive rehabilitation treatment followed by a telemedicine program on the motor, non-motor symptoms (pain, fatigue, anxiety, and depression), the self-perception of clinical change and Health-Related Quality of Life, and health care costs in patients with FMDs.

DETAILED DESCRIPTION:
Functional movement disorders (FMDs) are part of a broad spectrum of functional neurological disorders characterized by abnormal movements (gait, dystonia, and tremor), which are clinically incongruent with movement disorders caused by neurological disease and are significantly altered distraction or nonphysiologically maneuvers. FMDs have an incidence ranging from 4 to 12 per 100.000 population per year and a high prevalence (15-20%) in patients accessing neurological clinics. They are high disabling conditions characterized by long-term disability, poor quality of life, and economic impact on health and social care systems. Indeed, these patients experience disability and distress equivalent to those suffering from degenerative neurological diseases, such as Parkinson's Disease. Despite this, FMDs have been widely misunderstood, receiving little public and academic attention. Motor deficits, gait and balance disorders, and sensory manifestations are the most frequent symptoms and the leading cause of disability in patients with FMDs. They may occur in an isolated or combined manner, increasing the clinical complexity of these patients. Motor FMDs include functional poverty of movements, weakness, and slowness. Pain and fatigue are invalidating non-motor symptoms (NMSs) associated with FMDs. The pathophysiology of FMDs and their management remain largely unknown. The old assumption of psychological factors as the primary cause (psychogenic illness) has been abandoned due to the lack of evidence about their causal role. They have been removed from the diagnostic criteria described in the DSM-V and are considered risk factors.

Recent research findings suggest three key processes involved in the neurobiology of FMD: abnormal attentional focus, abnormal beliefs/expectations, and abnormalities in the sense of agency. Rehabilitation is essential in managing FMDs to improve function and quality of life in the context of a multidisciplinary team. Of note, patients with functional motor disorder may have much greater potential for recovery than health professionals often consider. However, three unmet needs remain crucial. Firstly, rehabilitation approaches are few and limited because empirical approaches mainly refer to clinical practice without following evidence-based consensus recommendations. Secondly, most existing studies are uncontrolled case series or crossover studies. Finally, adjuncts and innovations to improve access to specialist rehabilitation treatment by qualified professionals (i.e., tele/remote health and wearable technology) and monitor patients in the long-term have seldom been explored in patients with FMDs. The literature shows how these patients generally feel misunderstood and neglected by health professionals, becoming progressively more vulnerable. The connectivity of mobile devices with the internet ushered in technology platforms like telemedicine and wearable sensors, endowing hand-held devices with the ability to acquire and track data on physiologic systems (i.e., cardiovascular, gait) in the ecological setting at home and during the Activities of Daily Living. This introduced a new path for generating a new form of healthcare through the medical data acquisition by the individual, in real-time, in a real-world environment. Telemedicine overcomes the barrier of distance and time and provides access to patients having temporary and permanent disabilities for accurate diagnosis and rehabilitation prescription and delivery. To the best of our knowledge, no studies have been performed on the effectiveness of digital telerehabilitation on motor and non-motor outcomes and quality of life in patients with FMDs. A range of factors supports the implementation of digital telerehabilitation treatments in managing patients with FMDs.

Aims of the project Primary aim: To compare the effects of a telemedicine program on motor symptoms severity and duration in patients with FMDs.

Secondary aim: to compare the training effects on non-motor symptoms (pain, fatigue, anxiety, and depression), the self-perception of clinical change and Health-Related Quality of Life, and health care costs.

ELIGIBILITY:
Inclusion Criteria:

* a clinically definite diagnosis of FMDs based on Gupta and Lang diagnostic criteria with the presence of distractibility maneuvers and a demonstration of positive signs;
* the presence of 1 (isolated FMDs) or more clinical motor symptoms (combined FMDs), including weakness, tremor, jerks, dystonia, gait disorders, and parkinsonism;
* acceptable level of digital skills.

Exclusion Criteria:

* prominent dissociative seizures
* prominent cognitive and physical impairment that precludes signing the informed consent for participation in the study;
* unable or refuse to attend the consecutive 5-day rehabilitation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in the Simplified Functional Movement Disorders Rating Scale (S-FMDRS) score | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  Objective-rated validated scale to rate the duration and severity of functional motor symptoms (range: 0-54; higher = worse).

SECONDARY OUTCOMES:
Change in the Multidimensional Fatigue Inventory Scale (MFI-20) score | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It evaluates fatigue differentiating general, physical, reduced-activity, reduced-motivation, and mental fatigue (subscale range: 4-20; higher = worse).
Change in the Brief Pain Inventory (BPI) score | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It evaluates pain intensity (range: 0-40; higher = worse) and interference (range: 0-70; higher = worse).
Change in the Beck Depression Inventory (BDI-II) score | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It evaluates depression (range: 0-63; higher = worse).
Change in the Beck Anxiety Inventory (BAI) score | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It evaluates anxiety (range: 0-63; higher = worse).
Change in the 12-item Short-Form Health Survey (SF-12) score | before the intensive 5-day rehabilitation program (T0), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  The health-Related QoL will be evaluated by the Mental Health and Physical functioning of the 12-item Short-Form Health Survey (SF-12) (range: 0-100; higher = better)
Change in the Clinical Global Impression (CGI) score | the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  Self-rated perception of change will be assessed with the 7-point Clinical Global Impression (CGI) scale with scores from 1 (very much improved) to 7 (very much worse).
Change in the spatio-temporal gait parameters | before the intensive 5-day rehabilitation program (T0), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  Gait analysis will be used to collect gait speed (cm/s), cadence (step/min), and stride length (cm).
Change in the postural control assessment | before the intensive 5-day rehabilitation program (T0), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  An electronic monaxial stabilometric platform will be used to evaluate postural control.
Healthcare Services Volume ad-hoc questionnaire | before the intensive 5-day rehabilitation program (T0), and at 24 weeks (follow-up, T3)
  The number of the health services consulted six months before the intensive 5-day rehabilitation program will be retrospectively collected through an ad-hoc questionnaire. The same information will be prospectively collected during the study period (6 months).
Change in the Toronto Alexithymia Scale (TAS-20) score | before the intensive 5-day rehabilitation program (T0), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It evaluates the level of alexithymia (range: 20-100; higher = worse),
Number of direct Healthcare Costs consumption by an ad-hoc questionnaire | before the intensive 5-day rehabilitation program (T0), and 24 weeks (follow-up, T3)
  The number of examinations, medications, medical visits, hospital admissions, and Emergency Room visits performed before the intensive 5-day rehabilitation will be retrospectively collected through an ad-hoc questionnaire. The same information will be prospectively collected during the study period (6 months).
Number of days off. | before the intensive 5-day rehabilitation program (T0), after 12 weeks (at the end of the self-management plan, T2),and after 24 weeks (follow-up, T3)
  The number of days off for the patient.

OTHER OUTCOMES:
Number of drop-out | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  the number of dropouts before the end of treatment will be collected. The EG will report adverse events on the Digital Telemedicine platform, while the CG on the paper log.
Number of falls or events near falling. | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  The number of falls or events near falling will be collected on the on the Digital Telemedicine platform, while the CG on the paper log.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Schena, PhD, Study Director — Universita di Verona
Locations (1):
- USD Parkinson's Disease and Movement Disorders Unit, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez DL, Edwards MJ, Nielsen G, Kozlowska K, Hallett M, LaFrance WC Jr. Decade of progress in motor functional neurological disorder: continuing the momentum. J Neurol Neurosurg Psychiatry. 2021 Mar 15:jnnp-2020-323953. doi: 10.1136/jnnp-2020-323953. Online ahead of print. PMID 33722822
- [Background] Tinazzi M, Morgante F, Marcuzzo E, Erro R, Barone P, Ceravolo R, Mazzucchi S, Pilotto A, Padovani A, Romito LM, Eleopra R, Zappia M, Nicoletti A, Dallocchio C, Arbasino C, Bono F, Pascarella A, Demartini B, Gambini O, Modugno N, Olivola E, Di Stefano V, Albanese A, Ferrazzano G, Tessitore A, Zibetti M, Calandra-Buonaura G, Petracca M, Esposito M, Pisani A, Manganotti P, Stocchi F, Coletti Moja M, Antonini A, Defazio G, Geroin C. Clinical Correlates of Functional Motor Disorders: An Italian Multicenter Study. Mov Disord Clin Pract. 2020 Sep 22;7(8):920-929. doi: 10.1002/mdc3.13077. eCollection 2020 Nov. PMID 33163563
- [Background] Espay AJ, Aybek S, Carson A, Edwards MJ, Goldstein LH, Hallett M, LaFaver K, LaFrance WC Jr, Lang AE, Nicholson T, Nielsen G, Reuber M, Voon V, Stone J, Morgante F. Current Concepts in Diagnosis and Treatment of Functional Neurological Disorders. JAMA Neurol. 2018 Sep 1;75(9):1132-1141. doi: 10.1001/jamaneurol.2018.1264. PMID 29868890
- [Background] Nielsen G, Stone J, Matthews A, Brown M, Sparkes C, Farmer R, Masterton L, Duncan L, Winters A, Daniell L, Lumsden C, Carson A, David AS, Edwards M. Physiotherapy for functional motor disorders: a consensus recommendation. J Neurol Neurosurg Psychiatry. 2015 Oct;86(10):1113-9. doi: 10.1136/jnnp-2014-309255. Epub 2014 Nov 28. PMID 25433033
- [Background] Gupta A, Lang AE. Psychogenic movement disorders. Curr Opin Neurol. 2009 Aug;22(4):430-6. doi: 10.1097/WCO.0b013e32832dc169. PMID 19542886
- [Background] Gandolfi M, Riello M, Bellamoli V, Bombieri F, Geroin C, Di Vico IA, Tinazzi M. Motor and non-motor outcomes after a rehabilitation program for patients with Functional Motor Disorders: A prospective, observational cohort study. NeuroRehabilitation. 2021;48(3):305-314. doi: 10.3233/NRE-201617. PMID 33780378
- [Derived] Gandolfi M, Landi S, Sandri A, Di Vico IA, Geroin C, Menaspa Z, Maistri G, Fasoli M, Schena F, Tinazzi M, Leardini C. Clinical outcomes and economic impact of a digital telemedicine intervention in patients with functional motor disorders: a single-blind, randomised controlled trial. J Neurol Neurosurg Psychiatry. 2025 Dec 12;97(1):81-90. doi: 10.1136/jnnp-2025-336437. PMID 40912911